CLINICAL TRIAL: NCT02217787
Title: A Phase 1, Cross-over, Randomized, Single-dose Open Label Study To Determine The Effect Of Food On The Pharmacokinetics Of Orally Administered Pf-06372865 In Healthy Adult Subjects
Brief Title: Food Effect Study for PF-06372865
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7431008; 2014-002967-13 (EudraCT Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-15 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — PF-06372865

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fasted condition (Other)
  Interventions: Drug: PF-06372865
- fed condition (Other)
  Interventions: Drug: PF-06372865

INTERVENTIONS:
Drug: PF-06372865 — 7.5 mg as 3 x 2.5 mg tablets single dose
  Arms: fasted condition
Drug: PF-06372865 — 7.5 mg as 3 x 2.5 mg tablets single dose
  Arms: fed condition

SUMMARY:
This study has been designed to investigate the effect of high fat food on the pharmacokinetics of PF-06372865 when administered to healthy subjects as single oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs);

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Screening supine blood pressure > 140 mm Hg (systolic) or >90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Any condition possibly affecting drug absorption: current or recent (within one year) gastrointestinal disease; a history of malabsorption, esophageal reflux, irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn; or any surgical intervention (e.g., cholecysectomy) which would be expected to influence the absorption of drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | basline to 48 hours
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | basline to 48 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Concentration (Cmax) | basline to 48 hours
Time to Reach Maximum Observed Plasma Concentration (Tmax) | basline to 48 hours
Plasma Decay Half-Life (t1/2) | basline to 48 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

SECONDARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure | basline to 48 hours
  Value at time T minus value at baseline.
Change from Baseline in Diastolic Blood Pressure | basline to 48 hours
  Value at time T minus value at baseline.
Change from baseline in heart rate | basline to 48 hours
  value at time T minus value at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7431008&StudyName=Food%20effect%20study%20for%20PF-06372865%20